CLINICAL TRIAL: NCT04853394
Title: MASLIHAT Intervention for Tajik Male Migrants Who Inject Drugs
Brief Title: Tajik Migrant Health Education Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Prisma Research Center (Unknown)
Responsible Party: Principal Investigator, Mary Ellen Mackesy-Amiti, Research Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-0795; R01DA050464 (NIH)
Record Dates: First submitted 2021-04-16; First posted 2021-04-21 (Actual); Results first posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections; Hepatitis C; Risky Health Behavior; Risk Reduction Behavior
Keywords: injection drug use; migrant workers; risk behavior
MeSH Terms: conditions — HIV Infections; Hepatitis C; Health Risk Behaviors; Risk Reduction Behavior; Risk-Taking

STUDY DESIGN:
Intervention Model Description: cluster-randomized parallel groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MASLIHAT peer education (Experimental): A peer educator prevention intervention program consisting of five weekly 2-hour small group sessions.
  Interventions: Behavioral: MASLIHAT
- TANSIHAT health education (Sham Comparator): A health education program consisting of five weekly 2-hour sessions small group sessions.
  Interventions: Behavioral: TANSIHAT

INTERVENTIONS:
Behavioral: MASLIHAT — peer educator intervention
  Arms: MASLIHAT peer education
Behavioral: TANSIHAT — health education intervention
  Arms: TANSIHAT health education

SUMMARY:
This study will test the efficacy of a peer-education prevention intervention to reduce risky drug, alcohol, and sexual behaviors among male Tajik labor migrants who inject drugs (MWID) while working in Moscow. The peer educator intervention will be compared to a health education control intervention. Each intervention consists of 5 weekly 2-hour small group sessions. Follow-up assessments will be conducted at 3, 6, 9, and 12 months after the intervention. It is hypothesized that, compared to MWID who receive the health education control intervention, those who receive the peer educator intervention will have a greater reduction in the frequency of risk behaviors. Similar effects are expected for network members of intervention participants.

DETAILED DESCRIPTION:
The investigators will recruit male Tajik migrants who inject drugs from 12 different sites in Moscow, including bazaars and other work sites. In both study arms, the recruited men (index participants) will be required to recruit two eligible MWID peers for interviews prior to being interviewed themselves. Participants will be randomly assigned to either the peer educator intervention program or the health education intervention program. After peer-recruited network members are enrolled and interviewed, the index participant will participate in the peer educator training or the control group activities. All participants and recruited network members will then be followed and re-interviewed at 3-month intervals for one year to assess changes in risky drug, alcohol, and sexual behaviors due to intervention participation and through diffusion to network members. The investigators will also collect data from voluntary HIV and HCV testing conducted at 6 months (HCV only) and at 12 months (HIV and HCV) post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* adult Tajik man
* injected drugs in past 30 days
* living and working as migrant laborer in Moscow

Exclusion Criteria:

* does not intend to stay in Moscow for the next 12 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-10-19 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Mackesy-Amiti, Ph.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- PRISMA Research Center, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Yes
The final data will be shared by depositing it in a public data repository. The final dataset will include self-reported sociodemographic characteristics, HIV transmission knowledge and risk awareness, sexual partners and risk behavior, illicit drug use and injection risk behavior, prevention self-efficacy, and injection drug use network interactions at 5 time points, and HIV and HCV test results at 2 time points. No identifying information will be included in the final dataset.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be made available upon study completion.
Access Criteria: Access will be provided upon request with a description of the intended use.

REFERENCES:
- [Background] Mackesy-Amiti ME, Levy JA, Bahromov M, Jonbekov J, Luc CM. HIV and Hepatitis C Risk among Tajik Migrant Workers Who Inject Drugs in Moscow. Int J Environ Res Public Health. 2023 May 24;20(11):5937. doi: 10.3390/ijerph20115937. PMID 37297541
- [Background] Luc CM, Levy J, Bahromov M, Jonbekov J, Mackesy-Amiti ME. HIV knowledge, self-perception of HIV risk, and sexual risk behaviors among male Tajik labor migrants who inject drugs in Moscow. BMC Public Health. 2024 Jan 11;24(1):156. doi: 10.1186/s12889-023-17543-1. PMID 38212755
- [Result] Mackesy-Amiti ME, Bahromov M, Levy JA, Jonbekov J, Luc CM. Changes in risk behaviour following a network peer education intervention for HIV prevention among male Tajik migrants who inject drugs in Moscow: a cluster-randomized controlled trial. J Int AIDS Soc. 2024 Jul;27 Suppl 3(Suppl 3):e26310. doi: 10.1002/jia2.26310. PMID 39030891
- [Derived] Mackesy-Amiti ME, Levy JA, Luc CM, Jonbekov J. Peer education intervention reduced sexually transmitted infections among male Tajik labor migrants who inject drugs: results of a cluster-randomized controlled trial. BMC Public Health. 2025 Jun 10;25(1):2154. doi: 10.1186/s12889-025-23387-8. PMID 40495129
- [Derived] Mackesy-Amiti ME, Levy JA, Luc CM, Jonbekov J. Peer Education Intervention Reduced Sexually Transmitted Infections Among Male Tajik Labor Migrants Who Inject Drugs: Results of a Cluster-randomized Controlled Trial. medRxiv [Preprint]. 2025 May 1:2024.08.15.24312070. doi: 10.1101/2024.08.15.24312070. PMID 39185538
- See also: Open Science Framework Project page — https://osf.io/7g3yh/
- See also: Data files — https://osf.io/krjqs/?view_only=7c93ea8cf8384dce91b2b531000e63e3

RESULTS

PARTICIPANT FLOW:
Period: Baseline Interview
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Started | 210 | 210
Completed | 210 | 210
Not Completed | 0 | 0
Period: Intervention Sessions
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Started (Network member participated in interviews only) | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0
Period: Follow-up Interviews
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Started | 210 | 210
Completed | 188 | 195
Not Completed | 22 | 15
Not completed — Lost to Follow-up | 22 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education | Total
Number analyzed (Participants) | 210 | 210 | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 210 | 210 | 420
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (6.1) | 30.3 (6.3) | 30.0 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 210 | 210 | 420
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Tajik | 210 | 210 | 420
Region of Enrollment [Number; unit: participants]
  Russia | 210 | 210 | 420
Receptive syringe sharing [Count of Participants; unit: Participants] — injecting with a previously used syringe in the past 3 months
  Participants | 158 | 161 | 319
Condomless sex [Count of Participants; unit: Participants] — any condomless sex in the past 3 months
  Participants | 85 | 85 | 170
Binge alcohol use [Count of Participants; unit: Participants] — six or more drinks at a time at least once a month
  Participants | 45 | 43 | 88
Days of alcohol use past month [Mean (Standard Deviation); unit: days] | 5.2 (3.2) | 5.3 (3.4) | 5.3 (3.3)
HIV positive test result [Count of Participants; unit: Participants] — Population: Among participants with reported test results
  Participants
    number analyzed (Participants) | 207 | 206 | 413
    (all) | 19 | 9 | 28
Hepatitis C antibody positive test result [Count of Participants; unit: Participants] — Population: Among participants with reported test results
  Participants
    number analyzed (Participants) | 207 | 206 | 413
    (all) | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Syringe Sharing
Description: injected with a previously used syringe
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Number analyzed (Participants) | 210 | 210
Participants
  3-month follow-up | 16 | 167
  6-month follow-up | 15 | 175
  9-month follow-up | 22 | 163
  12-month follow-up | 36 | 163
Statistical Analysis 1: Comparison: MASLIHAT Peer Education vs TANSIHAT Health Education; Test type: Superiority; p < .01, Mixed Models Analysis; Mixed effects modified Poisson regression model with random intercepts for participant and network cluster; Risk Ratio (RR) = .33, 95% CI 2-sided [.21 to .51] — Effect of MASLIHAT vs. comparison TANSIHAT condition at 12-month follow-up

2. Primary Outcome: Sex Without Condom
Description: vaginal or anal sex without a condom in the past 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Number analyzed (Participants) | 210 | 210
Participants
  3-months | 27 | 77
  6-months | 25 | 91
  9-months | 25 | 86
  12-months | 26 | 93
Statistical Analysis 1: Comparison: MASLIHAT Peer Education vs TANSIHAT Health Education; Test type: Superiority; p = .01, Mixed Models Analysis; Mixed effects modified Poisson regression model with random intercepts for participant and network cluster; Risk Ratio (RR) = .67, 95% CI 2-sided [.46 to .97] — Effect of MASLIHAT vs. comparison TANSIHAT condition at 12-month follow-up

3. Primary Outcome: Alcohol Use
Description: Number of days drinking alcohol in past month
Time Frame: 30 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Number analyzed (Participants) | 210 | 210
days
  3-months | 4.5 (2.4) | 5.1 (2.8)
  6-months | 4.6 (2.3) | 5.2 (2.6)
  9-months | 5.6 (3.4) | 5.3 (2.6)
  12-months | 5.7 (2.3) | 6.1 (2.4)
Statistical Analysis 1: Comparison: MASLIHAT Peer Education vs TANSIHAT Health Education; Test type: Superiority; p = .01, Mixed Models Analysis; Mixed effects Poisson regression model with random intercepts for participant and network cluster; Risk Ratio (RR) = .86, 95% CI 2-sided [.77 to .95] — Effect of MASLIHAT vs. comparison TANSIHAT condition at 6-month follow-up
Statistical Analysis 2: Comparison: MASLIHAT Peer Education vs TANSIHAT Health Education; Test type: Superiority; p = .01, Mixed Models Analysis; Mixed effects Poisson regression model with random intercepts for participant and network cluster; Risk Ratio (RR) = 1.19, 95% CI 2-sided [.98 to 1.45] — Effect of MASLIHAT vs. comparison TANSIHAT condition at 12-month follow-up

4. Secondary Outcome: HIV Infection
Description: incident HIV infection
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Number analyzed (Participants) | 179 | 188
Participants | 0 | 0

5. Secondary Outcome: Hepatitis C Infection
Description: incident hepatitis C virus (HCV) infection
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Number analyzed (Participants) | 179 | 187
Participants | 3 | 3

6. Other Pre Specified Outcome: Injection Equipment Sharing
Description: used shared injection equipment
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
Number analyzed (Participants) | 210 | 210
Participants
  3-months | 16 | 168
  6-months | 16 | 170
  9-months | 15 | 160
  12-months | 15 | 164
Statistical Analysis 1: Comparison: MASLIHAT Peer Education vs TANSIHAT Health Education; Test type: Superiority; p = .01, Mixed Models Analysis; Mixed effects Poisson regression model with random intercepts for participant and network cluster; Risk Ratio (RR) = .12, 95% CI 2-sided [.07 to .19] — Effect of MASLIHAT vs. comparison TANSIHAT condition at 12-month follow-up

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | MASLIHAT Peer Education | TANSIHAT Health Education
All-Cause Mortality (participants affected / at risk) | 0/210 | 0/210
Serious Adverse Events (participants affected / at risk) | 0/210 | 0/210
Other Adverse Events (participants affected / at risk) | 3/210 | 3/210
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MASLIHAT Peer Education (N=210) | TANSIHAT Health Education (N=210)
hepatitis C infection (Infections and infestations) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/94/NCT04853394/Prot_SAP_000.pdf
  • Informed Consent Form: Index Participant (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04853394/ICF_001.pdf
  • Informed Consent Form: Network Participant (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/94/NCT04853394/ICF_002.pdf